CLINICAL TRIAL: NCT03609450
Title: Mindfulness Influences on Self-regulation: Mental and Physical Health Implications -- Integrating Mindfulness Into the Patient-Centered Medical Home (Phase 3)
Brief Title: Integrating Mindfulness Into the Patient-Centered Medical Home (Phase 3)
Acronym: MINDFUL-PC-3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1002/08/14_3; UH3AT009145 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Depression; Anxiety Disorders; Stress Related Disorder; Adjustment Disorders; Chronic Illness
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders; Chronic Disease | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Two arms, intervention and low-dose comparator, which are randomly assigned at the same time and are implemented in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training for Primary Care (Active Comparator): Mindfulness Training for Primary Care (MTPC) is a primary care adaptation that includes core common Mindfulness-Based Intervention (MBI) elements integrated with novel mindfulness-oriented behavior change elements into a format that is adaptable to delivery in primary care health centers.
  Interventions: Behavioral: Mindfulness Training for Primary Care
- Low-Dose Comparator (Other): Comparator arm: Participants receive a 60-minute introduction to mindfulness group plus referral to a list of community mindfulness resources such as private-pay community mindfulness classes, mobile mindfulness applications, books, and online recordings. These participants are added to a 6-month wait-list for a Cambridge Health Alliance mindfulness-based intervention group, but are allowed to receive behavioral, psychiatric, and medical treatments that are consistent with treatment as usual. All participants complete an action planning protocol during Week 7.
  Interventions: Behavioral: Low-Dose Comparator

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care — MTPC is a referral-based, insurance-reimbursable 8-week program delivered as group psychotherapy by Patient-Centered Medical Home-integrated behavioral clinicians or as an 8-week primary care group visit delivered by a primary care provider. MTPC groups are 2 hours for 8 weeks with a 7-hour weekend day of silent practice. MTPC emphasizes mindfulness-oriented skills for self-regulation, self-management of chronic illness, and health behavior change. All participants complete an action plan during Week 7. Participants are called every two weeks for the first eight weeks for 5-10 minute engagement calls which focus helping participants cultivate a relationship with study staff, giving participants a place to ask questions, and supporting participants in completing study visits.
  Arms: Mindfulness Training for Primary Care
Behavioral: Low-Dose Comparator — Participants in the low-dose comparator arm receive a 60-minute introduction to mindfulness. Participants are introduced to the definition(s) of mindfulness, brief mindfulness practices, and discussion. They are also given a list of leading community, online, print, and smartphone mindfulness resources. Participants are called every two weeks for the first eight weeks for 5-10 minute engagement calls which focus helping participants cultivate a relationship with study staff, giving participants a place to ask questions, and supporting participants in completing study visits.
  Arms: Low-Dose Comparator

SUMMARY:
This study compares the effectiveness of an 8-week mindfulness-based intervention (Mindfulness Training for Primary Care[MTPC]) vs. a low-dose mindfulness comparator on self-regulation targets, specifically the primary outcome of emotion regulation. Secondary outcomes include sustained attention/response inhibition and interoceptive awareness. A secondary analysis will investigate the extent to which these self-regulation targets mediate the impact of MTPC group on action plan initiation.

DETAILED DESCRIPTION:
The current Phase 3 comparative effectiveness randomized controlled trial examines impact of MTPC on specific mechanisms of change such as emotion regulation (primary outcome), interoceptive awareness and sustained attention/response inhibition (secondary outcomes). This study will also investigate the extent to which these self-regulation targets mediate the impact of MTPC group on action plan initiation. Participants randomized to 8-week MTPC are compared with participants randomized to a low-dose mindfulness comparator condition, in which they receive a 1-hour introduction to mindfulness with a referral to community mindfulness resources. Outcome assessments are conducted at baseline and study weeks 8-10. This study builds on the Phase 2 study, which demonstrated that Mindfulness Training for Primary Care enhanced chronic illness self-management action plan initiation among primary care patients receiving care in an urban, community, multi-cultural safety net healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Current CHA patient with an enrolled CHA primary care doctor.
2. CHA patients 18 years of age and older.
3. Able to tolerate and participate in interviews and engage in all procedures.
4. Able to give written consent in English OR willing and able to provide consent and complete assessments through a professional language translator when necessary.
5. Diagnosis eligible to be covered by insurance for group visits (e.g., anxiety disorder, depression, stress disorders including adjustment disorder related to chronic illness, pain, insomnia, etc.).
6. Must have access to a smartphone that is compatible with the activity tracker application.
7. Must be willing to use the smartphone application and/or wear a wristband device every day during the study collection periods
8. Must be able to fill out the study questionnaires daily on a computer or compatible mobile device.
9. Must be willing to attend the two computer task sessions.

Exclusion Criteria:

1. Any cognitive impairment that precludes informed consent.
2. Patients who, in the opinion of the Principal Investigator, pose an imminent risk of suicide or danger to self or others.
3. Likelihood of potential incarceration such as a conviction or pending charges that may potentially result in imprisonment.
4. Previous enrollment or randomization of treatment in the present study within the 12 months.
5. Behaviors that may cause disruption to a mindfulness group.
6. Patients with symptoms of psychosis, thought disorder, and/or severe mental illness, including schizophrenia, schizoaffective, bipolar disorder, or a current severe episode of major depressive disorder.
7. Refusal of insurance to cover group psychotherapy treatment may lead to exclusion from participation in groups.
8. Patients in their third trimester of pregnancy who foresee conflicts that preclude their commitment to completing all activities.
9. Patients with highly unstable medical problems that put them at a high risk of hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Difficulty in Emotion Regulation Scale (DERS) | Week 8
  The Difficulties in Emotion Regulation (DERS) Scale is a 36-item self-report scale designed to assess emotional dysregulation using a 5 point Likert scale. The scale assesses 6 aspects of emotional dysregulation: non-acceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Subscales are summed and a lower total score represents a better outcome.

SECONDARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Week 8
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness. The 6 point Likert scale (ranging from 0-6) assesses 8 aspects of interoceptive awareness: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Subscales are averaged, and a higher total score represents a better outcome.
Sustained Attention to Response Task (SART) | Week 8
  Participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer.
Action Plan Initiation Survey (APIS-5) | Weeks 8 - 10
  Patient self-reported Action Plan Initiation is based on two-item in the APIS-5 self-report survey in which patients are asked to list their action plan SMART goal, if they met the goal and how much control they had over meeting the goal. The main outcome is a single-item response determining whether they met or did not meet the goal using a 7-point Likert scale (ranging from 1-7) with scores >=5 representing self-reported initiation of the goal.
Hypothetical Delay Discounting Task (HDDT) | Week 8
  This is a brief delay discounting task performed on a computer that presents a series of 5 discrete choice questions between delayed larger reward and smaller sooner reward in dollars.
Heart Beat Detection Task (HBDT) | Week 8
  This is a behavioral measure of interoceptive awareness. Participants are asked to count their heartbeat during three varying time intervals ranging from 30 to 60 seconds. In parallel, individuals' heart-rate will be measured by Kardia Mobile technology.
Perceived Stress Scale (PSS-14) | Week 8
  The Perceived Stress Scale (PSS-14) (14 items) measures the degree to which situations in life are stressful. Items are designed to evaluate how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5 point Likert scale from 0 (Never) to 4 (Very often).
Five Facet Mindfulness Questionnaire (FFMQ) | Week 8
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item scale that examines five factors that represent aspects of the current empirical conception of mindfulness. These five facets include: "observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience." Participants rate their degree of agreement with each of the items on a Likert-type scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true), with higher scores indicating higher experience of mindfulness.
Self-Compassion Scale-Short Form (SCS-SF) | Week 8
  The short-form Self-Compassion Scale (SCS-SF) is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. The scale is scored on a 5 point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored.
Self-Efficacy for Managing Chronic Disease (SECD-6) | Week 8
  The Self-Efficacy for Managing Chronic Disease Scale (SECD-6) is a 6-item scale that is used to evaluate a participant's ability to self-manage care for a chronic disease. SECD-6 asks participants to rate their confidence in their own ability to do certain activities, on a scale from 1 (not at all confident) to 10 (totally confident).
Patient Reported Outcomes Measurement Information System - Anxiety Short Form (PROMIS-ASF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale used to assess patient-reported health status for anxiety. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always).
Patient Reported Outcomes Measurement Information System - Depression Short Form (PROMIS-DSF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Depression Short Form 8a (PROMIS-DSF) is an 8-item scale used to assess patient-reported health status for depression. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always).
Three Factor Eating Questionnaire -Revised 18 (TFEQ-R18) emotional eating subscale | Week 8
  The Three Factor Eating Questionnaire is an 18-item scale measuring eating behavior with 4-point Likert scale (1-4). The questionnaire refers to current dietary practice and measures three different aspects of eating-related behavior: cognitive restraint of eating (CR: 6 items), uncontrolled eating (UE: 9 items) and emotional eating (EE: 3 items). Each score ranges from 0 to 100, with higher score and this study is primarily investigating emotional and uncontrolled eating subscales.
  indicative of greater level in the eating behavior of interest.
Food, Activity, and Sleep Tracking (FAST) Questionnaire | Weeks 7-8
  The Food, Activity, and Sleep Tracking (FAST) is a questionnaire with responsive logic, including up to 45-items. The questionnaire assesses daily sleep behavior, daily activity and exercise, and daily nutritional intake, using validated items from the National Cancer Institute (ASA-24) and National Sleep Foundation Sleep diary. Responses to individual items will be tracked daily and increases in health-promoting activity and decreases in harmful behavior will represent a better outcome.
Mobile Device Accelerometer-Based Activity | Weeks 7-8
  Mobile device activity tracking with accelerometry, measuring overall activity, median daily activity count, and minutes of Moderate-to-Vigorous Physical Activity (MVPA)

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demarzo MM, Montero-Marin J, Cuijpers P, Zabaleta-del-Olmo E, Mahtani KR, Vellinga A, Vicens C, Lopez-del-Hoyo Y, Garcia-Campayo J. The Efficacy of Mindfulness-Based Interventions in Primary Care: A Meta-Analytic Review. Ann Fam Med. 2015 Nov;13(6):573-82. doi: 10.1370/afm.1863. PMID 26553897
- [Background] Loucks EB, Schuman-Olivier Z, Britton WB, Fresco DM, Desbordes G, Brewer JA, Fulwiler C. Mindfulness and Cardiovascular Disease Risk: State of the Evidence, Plausible Mechanisms, and Theoretical Framework. Curr Cardiol Rep. 2015 Dec;17(12):112. doi: 10.1007/s11886-015-0668-7. PMID 26482755
- [Background] Guendelman S, Medeiros S, Rampes H. Mindfulness and Emotion Regulation: Insights from Neurobiological, Psychological, and Clinical Studies. Front Psychol. 2017 Mar 6;8:220. doi: 10.3389/fpsyg.2017.00220. eCollection 2017. PMID 28321194
- [Background] Farb NA, Anderson AK, Segal ZV. The mindful brain and emotion regulation in mood disorders. Can J Psychiatry. 2012 Feb;57(2):70-7. doi: 10.1177/070674371205700203. PMID 22340146
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Mccubbin T, Dimidjian S, Kempe K, Glassey MS, Ross C, Beck A. Mindfulness-based stress reduction in an integrated care delivery system: one-year impacts on patient-centered outcomes and health care utilization. Perm J. 2014 Fall;18(4):4-9. doi: 10.7812/TPP/14-014. PMID 25662520
- [Background] Hallion LS, Steinman SA, Tolin DF, Diefenbach GJ. Psychometric Properties of the Difficulties in Emotion Regulation Scale (DERS) and Its Short Forms in Adults With Emotional Disorders. Front Psychol. 2018 Apr 19;9:539. doi: 10.3389/fpsyg.2018.00539. eCollection 2018. PMID 29725312
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Jha AP, Morrison AB, Dainer-Best J, Parker S, Rostrup N, Stanley EA. Minds "at attention": mindfulness training curbs attentional lapses in military cohorts. PLoS One. 2015 Feb 11;10(2):e0116889. doi: 10.1371/journal.pone.0116889. eCollection 2015. PMID 25671579
- [Background] Gawande R, To MN, Pine E, Griswold T, Creedon TB, Brunel A, Lozada A, Loucks EB, Schuman-Olivier Z. Mindfulness Training Enhances Self-Regulation and Facilitates Health Behavior Change for Primary Care Patients: a Randomized Controlled Trial. J Gen Intern Med. 2019 Feb;34(2):293-302. doi: 10.1007/s11606-018-4739-5. Epub 2018 Dec 3. PMID 30511291
- [Derived] Gawande R, Smith L, Comeau A, Creedon TB, Wilson CL, Griswold T, Cook BL, Loucks EB, Schuman-Olivier Z. Impact of warm mindfulness on emotion regulation: A randomized controlled effectiveness trial. Health Psychol. 2023 Oct;42(10):699-711. doi: 10.1037/hea0001303. Epub 2023 Jul 6. PMID 37410421

DOCUMENTS (1):
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03609450/ICF_001.pdf